CLINICAL TRIAL: NCT03342755
Title: Evaluation of STaged Endovascular Aneurysm Repair in the Management of Thoracoabdominal Pathology by Means of Branched and Fenestrated Devices.(STEAR)
Acronym: STEAR
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, MD, IRCCS San Raffaele
Other Study IDs: STEAR/33/OSR
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Thoracoabdominal Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to analyzing the impact of the staged endovascular treatment (divided into two or more distinct procedures) of thoracoabdominal aneurysmatic pathology on short and medium term, technical and clinical outcomes and on the possible benefits or complications associated with this approach.

DETAILED DESCRIPTION:
Since the development of custom-made fenestrated and branched endografts a novel therapeutic option for the management of thoracoabdominal aortic aneurysms was made accessible. In order to achieve complete aneurysm exclusion more than one endovascular graft is usually needed according to device characteristics and aneurysm extent. Usually a straight tube graft is initially placed in the proximal descending aorta, followed by a custom-made device for the visceral abdominal aorta, and completed with a bifurcated infrarenal graft landing at the level of the common iliac arteries. Many variations are available according to patient anatomy, pathology, and previous aortic surgeries.

The different components required can be deployed in the patient in one setting (i.e. single-stage endovascular repair) or across more than one surgeries (i.e. multi-stage endovascular repair), depending on procedural needs and surgeon choice. According to limited reported series the latter option seems to be associated to better clinical outcomes both in terms of spinal cord ischemia and overall survival.

In addition to the number, type and order of stages required for patient treatment, primary and secondary end-points are the evaluation of the short-term (6 months) and mid-term (5 years) outcomes as illustrated in the Society for Vascular Surgery reporting standards for TEVAR.

The investigators review a prospectively compiled Microsoft Office Excel database with the procedural details of the 47 patients treated at our Institution between October 2013 and October 2017 by means of total endovascular thoracoabdominal aortic aneurysm repair and of those of the next 50 patients which will be treated until December 2020. All patients will be recorded together with their characteristics and number and type of stages required for treatment completion.

All enrolled patients will be contact yearly by phone, in addition to standard follow-up imaging, to confirm persistence of technical and clinical success and to evaluate the eventual onset of any treatment related complication or disease evolution Possible stage types will be differentiated as: proximal thoracic component (TEVAR), visceral component (Custom-Made), bifurcated component (EVAR), iliac extensions, iliac branch devices.

All but the visceral component may or may not be present in each patient depending on the aneurysm extension and previous aortic surgery.

All the assessed variables will be prospectively recorded in a Microsoft Office Excel database together with patients' data.

All patients involved in the retrospective part of the study have already signed informed consent for data collection and analysis at hospital admission.

The 50 patients that will be enrolled until December 2020 will also sign an "ad hoc" consents, specific for this study.

Sensitive patient information will not be available during data analysis. The clinical study will be carried out according to the ethical principles of the Declaration of Helsinki and following the active regulations on observational studies.

Participation in the study does not involve ethical implications as the patients in the study will be subjected to the standard procedures commonly used to treat the pathology from which they are affected. The investigators just want to store participant' s data in anonymous database.

Patients characteristics, procedural data, technical and clinical outcomes, and follow-up data will be analyzed on Wizard Statistics software to investigate the presence of statistically significant correlations among the identified variables.

The extracted data will be the property of the investigator and San Raffaele Hospital, and their relevant clinical and procedural implications will be submitted for publication in peer-reviewed scientific journals focused on the field of vascular and endovascular surgery. Also in these works the data will be reported anonymously.

ELIGIBILITY:
Inclusion Criteria:

patient with ≥ 18 years of age, undergoing total endovascular treatment of thoracoabdominal pathology (single-stage or multi-stage endovascular repair) at San Raffaele Hospital in between October 2013 and December 2020.

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing total endovascular treatment of thoracoabdominal pathology (single-stage or multi-stage endovascular repair) at San Raffaele Hospital in between October 2013 and December 2020
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Prevention of rupture of aortic aneurysm or other aortic pathology | between October 2013 and December 2020
Prevention of death from aneurysm rupture or other aortic pathology (including end-organ ischemia) | between October 2013 and December 2020
Prevention of death associated with primary or secondary treatment of the original aortic pathology, including operative or endovascular intervention for rupture, dissection, or end-organ ischemia | between October 2013 and December 2020

SECONDARY OUTCOMES:
New, expanding, or progressing: aneurysm, dissection, ulceration, or hematoma | between October 2013 and December 2020
Device migration,degradation (eg, stent fracture, fabric erosion); | between October 2013 and December 2020
Endoleak presence (for aneurysm),Endoleak requiring intervention | between October 2013 and December 2020

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Callaghan A, Mastracci TM, Eagleton MJ. Staged endovascular repair of thoracoabdominal aortic aneurysms limits incidence and severity of spinal cord ischemia. J Vasc Surg. 2015 Feb;61(2):347-354.e1. doi: 10.1016/j.jvs.2014.09.011. Epub 2014 Oct 23. PMID 25449006
- [Background] Chuter TA, Rapp JH, Hiramoto JS, Schneider DB, Howell B, Reilly LM. Endovascular treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2008 Jan;47(1):6-16. doi: 10.1016/j.jvs.2007.08.032. Epub 2007 Nov 5. PMID 17980540
- [Background] Fillinger MF, Greenberg RK, McKinsey JF, Chaikof EL; Society for Vascular Surgery Ad Hoc Committee on TEVAR Reporting Standards. Reporting standards for thoracic endovascular aortic repair (TEVAR). J Vasc Surg. 2010 Oct;52(4):1022-33, 1033.e15. doi: 10.1016/j.jvs.2010.07.008. No abstract available. PMID 20888533